CLINICAL TRIAL: NCT03404453
Title: Difficult Airway Prediction in Paediatric Anaesthesia:Prospective Observational Trial
Brief Title: Difficult Airway Prediction in Paediatric Anaesthesia
Acronym: Diffair
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, doc.MD.Ph.D, Brno University Hospital
Other Study IDs: KDAR FN Brno Airway 2018
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Difficult Airway
Keywords: Airway prediction; Difficult airway

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paediatric patients at preanaesthetic visi: Difficult airway incidence and prediction:Paediatric patients at preanaesthetic visit scheduled for surgery under general anaesthesia
  Interventions: Diagnostic Test: Difficult airway incidence and prediction

INTERVENTIONS:
Diagnostic Test: Difficult airway incidence and prediction — Paediatric patients scheduled for surgery under general anaesthesia will be examined and a set up of airway prediction tests will be performed to predict the possibility of difficult airway

SUMMARY:
The incidence of difficult airway in paediatric population is up-to date not well described. Difficult airway is connected with significant airway-related morbidity and mortality. The majority of difficult airway in paediatric patients should be predictable. The aim of the study is to evaluate the incidence of difficult airway in paediatric patients scheduled for surgery under general anaesthesia and to test the predictability of the set of prediction tests to reveal the patients with high risk of difficult airway.

DETAILED DESCRIPTION:
At the preanaesthetic visit the paediatric patients will be examined for difficult airway. The Mallampati score, interincisor garp, cervical spine mobility, upper lip bite test and thyromental distance will be measured. The distances will be measured in centimeters and the width of the distal part of the third finger will be measured to obtain the distance according to the patients fingers. The airway management plan will be defined and the incidence of the difficult airway (difficult face mask ventilation - two hand, two operators, desaturation, difficult intubation - Cormack-Leehane 3-4, intubation on 3 and more attempts, difficult laryngeal mask insertion and the incidence of cannot intubate cannot ventilate scenario will be evaluated. The predictability of the test for difficult airway prediction (Cormack-Leehane 3-4, cannot-intubate - cannot ventilate scenario, difficult mask ventilation) will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

- All paediatric patients scheduled for surgery under general anaesthesia On the preanaesthetic examination

Exclusion Criteria:

- Airway already secured by tracheostomy Surgery without securing the airway

Ages: 28 Days to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: Paediatric patients at the preanaesthetic examination, scheduled for surgery under general anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of difficult airway in paediatric patients under general anaesthesia | during anaesthesia induction
  The incidence of the difficult airway will be evaluated by the anaesthesiologist in the operating room. Difficult airway will be considered as difficult face mask ventilation, difficult intubation (Cormack-Leehane 3 and 4, intubation at 3 and over 3rd attempt), difficult laryngeal mask insertion (more than 2 attempts) and the presence of the cannot intubate - cannot ventilate scenario.

SECONDARY OUTCOMES:
Predictability of difficult airway | during anaesthesia induction
  At the preanaesthetic examination a set of difficult airway prediction tests will be performed and the predictability of difficult airway will be evaluated by the statistical analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Brno University Hospital, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided